CLINICAL TRIAL: NCT04063605
Title: The Effect of Clinical Pilates Training on Balance and Postural Control of People With Parkinson's Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University of Lefke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ÜEK/32/02/03/1819/01; ÜEK/32/02/03/1819/01 (Other: European University of Lefke)
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: 2 groups will receive different exercise program for 8 weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Pilates (Experimental): Participants in this group will receive twice a week, total 8 weeks of clinical pilates exercise program. Each session will take 45 minutes.
  Interventions: Other: Clinical Pilates
- Classic Physiotherapy (Active Comparator): Participants in this group will receive twice a week, total 8 weeks of classic physiotherapy exercise program. Each session will take 45 minutes.
  Interventions: Other: Classic Physiotherapy

INTERVENTIONS:
Other: Clinical Pilates — This exercise model focus on the awareness of the neutral position of the spine and strengthen the deep postural muscles of the spine. Training of trunk muscles is emphasized and trunk stabilization is achieved and more difficult activities are initiated and thus, body awareness is improved. There are general principles to be followed during exercises. These; The principle of concentration is respiration, central focus, control, stability and isolation. These principles are achieved by simultaneous muscle activation of muscles responsible for trunk stabilization (multifidus, diaphragm, transversus abdominis and pelvic floor muscles). In order for an exercise to become a clinical pilates exercise, trunk stabilization must be ensured and breath control should be established in each exercise.
  Arms: Clinical Pilates
Other: Classic Physiotherapy — This exercise program will include strengthening, stretching, posture exercises, balance and gait exercises. Aim is to improve muscle strength and prevent shortness of muscles. Also, balance and gait exercise aim to improve walking capacity.
  Arms: Classic Physiotherapy

SUMMARY:
Many studies showed that clinical pilates exercises has positive effects on static and dynamic balance of different populations. It was suggested that this type of exercise reduce the risk of falls and physical damage. It also helps prevention of kyphotic posture. Parkinson's patients have both balance and postural problems but no study investigated the effect of clinical pilates exercises for this population. The aim of this study is to investigate the effects of clinical pilates exercise program on postural control and balance in individuals with Parkinson's disease.

DETAILED DESCRIPTION:
The patients will be randomly assigned into two groups: Clinical Pilates (CP) Group and Classic Physiotherapy (CF) Group. Both groups will be treated for 8 weeks. The evaluation of the patients will be done before the beginning of exercise program and will be repeated at the end. Static balance of patients will be evaluated with Single Leg Stance Test and Tandem Stance Test, dynamic balance with Functional Reach Test (FRT) and 30 second Chair Stand Test. Postural control and balance will also be evaluated with Berg Balance Scale and functional capacity by Timed Up and Go Test. Symptom severity and treatment complications of the patients will be evaluated with United Parkinson's Disease Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

* Stage 2-3 of Modified Hoehn & Yahr Scale
* 26 or> 26 points from the Mini Mental test
* Having at least 2 years Parkinson Disease

Exclusion Criteria:

* Serious mental and psychological disorder
* Significant musculoskeletal disorders
* Lower extremity deformation
* Having another neurological disease
* Drug or dose change during treatment

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
One leg stance test | 5 minutes
  This test is used to measure balance and standing ability and gives an idea about the individual's ability to balance and the risk of falling. Test measures how many seconds the patient can stand on one leg.
Tandem stance test | 5 minutes
  It is a test that evaluates the static balance by narrowing the ground contact area. The heel of one foot is adjusted to the end of the other foot. Patient is asked to try to stand without loss of balance and the time is recorded in seconds.
Functional reach test | 5 minutes
  A balance test designed to measure stability limits. The patient is asked to raise the dominant arm 90 ° and place it at the shoulder level and extend as far as it can go forward, without loss of movement or balance in the feet. Reduced ability to reach indicates an increased risk of falling in the future.
Sit-to-stand test | 5 minutes
  This test evaluates the patient's sit-up activity, lower extremity strength and dynamic balance. The patient's number of sitting and getting up within 30 seconds gives the test score.
Timed-up and Go test | 5 minutes
  When the command is given, the patient gets up from a normal chair, walks 3 meters, turns and walks back to the chair and sits down. The time starts when the command is given and ends when the person sits back in the chair.
Berg Balance Scale | 15 minutes
  This test is used to measure a person's static and dynamic balance performance. It is effective in assessing postural control and predicting the risk of falling. It is a 14-item test that uses 0 to 4 sequential scoring for each item. The total score range is from 0 to 56 and a higher score indicates a better balance.

CONTACTS AND LOCATIONS:
Overall Officials: Beliz Belgen Kaygisiz, PT, PhD, Principal Investigator — European University of Lefke
Locations (1):
- European University of Lefke, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- [Derived] Coban F, Belgen Kaygisiz B, Selcuk F. Effect of clinical Pilates training on balance and postural control in patients with Parkinson's disease: a randomized controlled trial. J Comp Eff Res. 2021 Dec;10(18):1373-1383. doi: 10.2217/cer-2021-0091. Epub 2021 Nov 2. PMID 34726472